CLINICAL TRIAL: NCT02739295
Title: Evaluation of G-CSF as a Treatment of Toxic Epidermal Necrolysis
Brief Title: G-CSF in the Treatment of Toxic Epidermal Necrolysis
Acronym: NeupoNET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Anne-Françoise Rousseau, MD, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L002
Record Dates: First submitted 2016-04-04; First posted 2016-04-15 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2023-06

CONDITIONS: Stevens - Johnson Syndrome
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — Filgrastim; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-CSF (Experimental): An intravenous dose of 5 microg/kg of G-CSF (Neupogen) will be administered daily, from admission (day 0) to day 4.
  Interventions: Drug: recombinant granulocyte - colony stimulating factor
- Placebo (Placebo Comparator): An intravenous dose of 5 ml of NaCl 0.9% will be administered daily, from admission (day 0) to day 4.
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: recombinant granulocyte - colony stimulating factor
  Other Names: Neupogen (Amgen)
  Arms: G-CSF
Drug: NaCl 0.9%
  Arms: Placebo

SUMMARY:
NeupoNET aims to evaluate interest of G-CSF in the treatment of Toxic Epidermal necrolysis. This is a prospective randomized controlled trial.

Patients will be allocated in a treatment group (receiving an injection of 5 microg/kg/d of G-CSF during 5 consecutive days) or in a placebo group. Patients will be randomized at admission and will be followed until 3 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Toxic epidermal necrolysis with SCORTEN 1 to 5 at admission

Exclusion Criteria:

* Toxic epidermal necrolysis with SCORTEN 6 or 7 at admission
* Hypercoagulable state
* Cardiac or peripheral arterial disease
* Active malignancy
* Myelodysplastic syndrome or hematological malignancy
* Fructose intolerance
* Pregnancy
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Time for healing | From date of randomization until the date of complete healing, assessed up to 30 days.
  Time for complete cutaneous healing, considered as healing of 90% of the body surface area
Immunohistology: Changes in immunohistologic typing (MAC 387, CD15, CD68, CD45Ro, fact XIIIa) | At admission and at day 5
  Changes in immunohistologic typing (MAC 387, CD15, CD68, CD45Ro, fact XIIIa)
Biological data: Neutrophilic count | Every day during the 14th first days
  Neutrophilic count

SECONDARY OUTCOMES:
Biological data: WBC count | 3 months after discharge
  WBC count
Biological data: WBC formula | 3 months after discharge
  WBC formula

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Burn Centre of the University Hospital of Liège, Liège
  - IMTR Burn Centre, Loverval

IPD SHARING:
Plan to Share IPD: No